CLINICAL TRIAL: NCT04788771
Title: Comparison of Tracheal Intubation and Laryngeal Mask Airway in Laparoscopic Total Extraperitoneal (TEP) Repair in Patients With Unilateral Inguinal Hernia
Brief Title: Comparison of Tracheal Intubation vs Laryngeal Mask Airway in Laparoscopic Total Extraperitoneal Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Turgut Donmez, Bakirkoy EAH, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BakirkoyEAH LMA
Record Dates: First submitted 2021-03-05; First posted 2021-03-09 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Lung Functions; Pain Score
MeSH Terms: interventions — Intubation, Intratracheal

STUDY DESIGN:
Intervention Model Description: Tracheal intubation
Who Masked: Investigator
Masking Description: laryngeal mask airway
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tracheal intubation in laparoscopic extraperitoneal hernia repair (Sham Comparator): Tracheal intubation in laparoscopic extraperitoneal hernia repair
  Interventions: Procedure: Tracheal intubation in laparoscopic extraperitoneal hernia repair
- laryngeal mask airway in laparoscopic extraperitoneal hernia repair (Active Comparator): laryngeal mask airway in laparoscopic extraperitoneal hernia repair
  Interventions: Procedure: Tracheal intubation in laparoscopic extraperitoneal hernia repair

INTERVENTIONS:
Procedure: Tracheal intubation in laparoscopic extraperitoneal hernia repair — laryngeal mask airway in laparoscopic extraperitoneal hernia repair

SUMMARY:
Patient comfort and satisfaction of inguinal hernia repairs can be affected by the anesthesia technique chosen in addition to the surgical method. In our study, we aimed to compare the anesthesia method used in patients during laparoscopic total extraperitoneal hernia repair, which is a minimally invasive method.It was planned to evaluate the patients' quality of life, pain conditions, additional medical support needs for pain, length of hospital stay, duration of surgery, complications during and after surgery and recurrence rates.In addition, it was planned to compare the effects of the anesthesia method used on the lung capacity of the patients. The most important achievement of the study will be to show that laparoscopic hernia repair, which is frequently performed by intubation, can be performed safely with the Laryngeal mask.

DETAILED DESCRIPTION:
The study was designed as a prospective randomized study, and a total of 100 patients were planned to be evaluated. Laparoscopic total extraperitoneal hernia repair will be performed by anesthesia with laryngeal mask and treceal intubation. Patients with a lariyngeal mask will be named as "group 1", and patients who undergo tracheal intubation will be named as "group 2".

Patients diagnosed with inguinal hernia radiologically and diagnosed with ultrasound will be operated. Patients between the ages of 18 and 75 years will be included in the study. Patients with relapse will be excluded. All patients will be evaluated for preoperative anesthesia and their suitability for laryngeal mask or tracheal intubation will be examined. Patients considered unsuitable for anyone will not be included in the study.

All patients will be explained in two methods before surgery and their patients will be randomized. Randomization will be done on the website www.randomizer.org. All patients will be entered on the website by numbering and the method chosen by the website will be applied according to the order of arrival.

Patients will be placed in the supine position under operating room conditions and anesthesia will be appropriate. After anesthesia, the surgical procedure will begin. The first incision time will be accepted as the surgery start time, and the end time of skin suturization will be recorded as the end of the surgery.

VAS scores of the patients at the 1st, 2nd, 4th, 6th and 12th hours after surgery will be learned and recorded by the service nurses. Additional medical needs of patients due to pain will be recorded.

Demographic data and additional diseases of the patients will be recorded. Operation times, hospitalization times, wound infections, seroma, scrotal edema and pain scores will be recorded. Complications developed during the operation will be recorded. After surgery, patients' nausea, vomiting, headache, shoulder pain and pain scores will be compared. Patients will be called to the general surgery outpatient clinic in the first week, first month, third month, and sixth month after the operation.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of unilateral inguinal hernia

Exclusion Criteria:

Clinical diagnosis of incarcerated inguinal hernia Clinical diagnosis of inguinal hernia with pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
VAS score | postoperative 1th hour vas score
  Evaluation of postoperative 1th hour pain score with VAS scale
Anatomical delineation: satisfactory (n)(%) | up to 2 hour
  Surgeon's evaluation at the end of the operation

SECONDARY OUTCOMES:
Sore throat | up to 2 hour
  sore throat that develops after surgery
Hoarsaness and dysphonia | up to 2 hour
  Hoarsaness and dysphonia develops after surgery
seroma | up to 30 day
  postoperative seroma
scrotal edema | up to 30 day
  postoperatif scrotal edema
ventilation time | up to 2 hour
  ventilation time during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Turgut Donmez, Principal Investigator — Bakırkoy Dr. Sadi Konuk Training and Research Hospital
Locations (1):
- Bakirkoy Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nevescanin A, Vickov J, Elezovic Baloevic S, Pogorelic Z. Laryngeal Mask Airway Versus Tracheal Intubation for Laparoscopic Hernia Repair in Children: Analysis of Respiratory Complications. J Laparoendosc Adv Surg Tech A. 2020 Jan;30(1):76-80. doi: 10.1089/lap.2019.0382. Epub 2019 Oct 15. PMID 31613680
- [Result] Nagahisa Y, Hashida K, Matsumoto R, Kawashima R, Okabe M, Kawamoto K. A randomized clinical study on postoperative pain comparing between the supraglottic airway device and endotracheal tubing in transabdominal preperitoneal repair (TAPP). Hernia. 2017 Jun;21(3):391-396. doi: 10.1007/s10029-017-1586-y. Epub 2017 Feb 13. PMID 28194529